CLINICAL TRIAL: NCT07352371
Title: Metaphors to Enhance Antibiotic Appropriate Use Knowledge and Behaviours to Reduce Educational Disparities Among Chinese Parents: A Survey-experimental Study
Brief Title: Metaphors to Enhance Antibiotic Appropriate Use Knowledge and Behaviours to Reduce Educational Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Yan (Other)
Collaborators: Hangzhou Normal University (Other)
Responsible Party: Sponsor-Investigator, Bo Yan, Dr., Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZGL202403-3; 72004194 (Other Grant/Funding Number: Natural Science Foundation of China)
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Antimicrobial Resistance
Keywords: metaphor; antimicrobial resistance; antibiotic use behaviour; equity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study is double-blinded, meaning that both the subjects and the researchers are unaware of the group assignments. The randomization of groups is conducted using Wenjuanxing (a survey tool). However, blinding is not implemented during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metaphorical messages group (Experimental): The metaphorical messages, by contrast, were crafted to be more accessible, drawing on familiar daily-life analogies derived from our prior qualitative research. We created three specific pairs: the first explained mechanisms of AMR, comparing resistant bacteria to pesticide-resistant insects. The second addressed environmental contamination by likening antibiotics to mercury batteries. The third used the analogy of "organic" food to convey the concept of antibiotic-free animal foods.
  Interventions: Behavioral: metaphorical messages
- conventional messages group (Placebo Comparator): The conventional messages were adapted from formal health communication sources, such as the World Health Organization and the Chinese National Health Commission, and retained the technical tone typical of official health education materials (China NHC, 2010; He, 2018; WHO, 2022).
  Interventions: Behavioral: conventional messages

INTERVENTIONS:
Behavioral: metaphorical messages — We created three specific pairs: the first explained mechanisms of AMR, comparing resistant bacteria to pesticide-resistant insects. The second addressed environmental contamination by likening antibiotics to mercury batteries. The third used the analogy of "organic" food to convey the concept of antibiotic-free animal foods. All metaphorical messages were reviewed by a panel of experts in public health, clinical microbiology, health communication, and health education to ensure factual consistency and clarity.
  Arms: metaphorical messages group
Behavioral: conventional messages — The conventional messages were adapted from formal health communication sources, such as the World Health Organization and the Chinese National Health Commission, and retained the technical tone typical of official health education materials (China NHC, 2010; He, 2018; WHO, 2022).
  Arms: conventional messages group

SUMMARY:
A randomized controlled survey experiment was conducted from October to November 2024 to assess the effectiveness of metaphor-based health education in improving Chinese parents' knowledge and behavioural intentions regarding appropriate antibiotic use. A total of 866 parents from two Chinese provinces were randomly assigned to either a metaphorical message group (n = 432) or a conventional message group (n = 434). Metaphors included comparing antimicrobial resistance (AMR) to insect resistance to pesticides, improper antibiotic disposal to mercury battery pollution, and antibiotic-free foods to organic foods. Outcomes measured were AMR knowledge, willingness to pay (WTP) for antibiotic-free foods, and proper antibiotic disposal intention.

DETAILED DESCRIPTION:
To assess the influence of metaphorical and conventional health education messages on the AMR-related knowledge and behavioural intentions of rural and urban residents, the investigators conducted a survey experimental study across two provinces in China. Prior to receiving any health education message, the respondents completed questions on AMR-related knowledge, behaviours, and behavioural intentions. Subsequently, participants were randomly assigned to read either metaphorical or conventional health education messages. Following the reading of assigned message, the respondents once again completed the questions on AMR-related knowledge and behavioural intentions.

ELIGIBILITY:
Inclusion Criteria:

* adult child parent, willing to participate

Exclusion Criteria:

* declining to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
knowledge | Immediately after the 30-second message exposure.
  Three items were summed to form the AMR-related knowledge scale. This scale was assessed by asking respondents to judge the correctness of the following statements before and after their first exposure to health education message: (1) Does antimicrobial resistance imply that bacteria are becoming increasingly difficult to kill with antibiotics? (2) Dose overuse of antibiotics lead to antimicrobial resistance? (3) Can antimicrobial resistant be transmitted between people?
Willingness to pay for antibiotic-free animal food | Immediately after the 30-second message exposure.
  Respondents were asked whether they were willing to pay a higher price for antibiotic-free animal foods compared to regular animal- foods. Their answers were dichotomized into "Yes" and "No/Not Sure".
antibiotic disposal intention | Immediately after the 30-second message exposure.
  To evaluate antibiotic disposal practices, participants were asked to recall how they had handled expired or unused antibiotic prior to receiving a third exposure to health education message.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Available on request.